CLINICAL TRIAL: NCT00020826
Title: An International Field Study Of The Reliability And Validity Of The EORTC QLQ-C30 And A Disease-Specific Questionnaire Module (The QLQ-STO22) In Assessing The Quality Of Life Of Patients With Gastric Cancer
Brief Title: Assessing Quality of Life of Patients With Stomach Cancer
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-15001-40003; EORTC-15001 (Other: EORTC); EORTC-40003 (Other: EORTC)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Gastric Cancer
Keywords: adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gastric adenocarcinoma: No protocol specific interventions. Both palliative or curative treatment allowed.
  Interventions: Other: quality-of-life assessment

INTERVENTIONS:
Other: quality-of-life assessment — QLQ-C30 questionnaire administered. STO22 questionnaire administered.
  Other Names: QLQ-C30 questionnaire administered.; STO22 questionnaire administered.

SUMMARY:
RATIONALE: Assessing quality of life in patients who are undergoing cancer treatment may help determine the effect of treatment on these patients.

PURPOSE: Clinical trial to study the effectiveness of a quality of life assessment in patients who are receiving treatment for stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the scale structure, reliability, and validity of the tumor-specific questionnaire, QLQ-STO22, in assessing the quality of life of patients with gastric cancer.
* Determine the questionnaire's sensitivity to change in clinical health status in these patients.

OUTLINE: Patients are stratified according to type of treatment (potentially curative vs potentially palliative), disease stage (local and locoregional vs metastatic), Karnofsky performance status (less than 80% vs more than 80%), and initial weight gain (none vs less than 10% of total body weight vs 10% or more of total body weight).

* Curatively Treated Group: Quality of life is assessed at 4 weeks prior to surgery and 3 months after surgery in patients receiving total or partial gastrectomy with curative intent; at 4 weeks prior to chemotherapy and/or radiotherapy, 4 weeks prior to surgery, and 3 months after surgery in patients receiving neoadjuvant chemotherapy and/or radiotherapy followed by total or partial gastrectomy with curative intent; at 4 weeks prior to chemotherapy and/or radiotherapy and 6 weeks after completion of therapy in patients receiving adjuvant chemotherapy and/or radiotherapy following total or partial gastrectomy; and at 4 weeks prior to therapy and 3 months after completion of therapy in patients receiving endoscopic mucosal resection or laparoscopic wedge resection.
* Palliatively Treated Group: Quality of life is assessed at 3 weeks prior to palliative therapy and 4 weeks after beginning palliative therapy.

PROJECTED ACCRUAL: Approximately 220 patients (110 per group) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric adenocarcinoma
* Patients treated with curative intent according to one of the following criteria:

  * Plan to undergo total or partial gastrectomy with curative intent
  * Plan to receive neoadjuvant chemotherapy and/or radiotherapy followed by total or partial gastrectomy with curative intent
  * Prior total or partial gastrectomy with curative intent and currently receiving adjuvant chemotherapy and/or radiotherapy
  * Prior endoscopic mucosal resection or laparoscopic wedge resection of early gastric cancer OR
* Patients with initial diagnosis of gastric cancer or recurrent disease with plans to receive one of the following therapies with palliative intent:

  * Total or partial gastrectomy or bypass procedure
  * Endoscopic procedure (e.g., stent insertion)
  * Chemotherapy and/or radiotherapy
  * Supportive measures only
* No concurrent enrollment on other quality of life study that would interfere with this study
* Not previously enrolled on this study

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Any performance status

Life expectancy:

* At least 2 months for patients treated with curative intent
* At least 4 weeks for patients treated with palliative intent

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent malignancies except basal cell carcinoma of the skin
* No mental impairment that would preclude completion of questionnaire
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be composed of a consecutive series of patients with gastric cancer meeting the eligibility criteria in each participating centre. The definition of gastric cancer is adenocarcinoma of the stomach, and includes all tumours of the fundus, body and antrum, linitis plastica and tumours of the cardia that infiltrate the gastro-oesophageal junction and distal oesophagus from below; classified as type III according to Siewert (1998. The study sample will be stratified by treatment - potentially curative and purely palliative.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2001-04; Primary Completion 2003-05 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
psychometric validity of the STO22 module | The EORTC QLQ-C30 and the gastric cancer module (QLQ-STO22) will be prospectively administered once before and once after primary treatment.
  Quality of life scores will be evaluated for psychometric validity by:
  * Scale structure using multi-trait scaling analysis
  * Reliability using tests of internal consistency
  * Test-retest reliability in patients recruited in the UK
  * Validity using inter-scale correlations and known group comparisons
  * Sensitivity to change using two measurements of Quality of Life and ANOVA to look for the significance of changes in quality of life scores as a function of observed changes in clinical status over time.

SECONDARY OUTCOMES:
debriefing questionnaire information | at baseline
  Patients will be asked to complete a short debriefing questionnaire covering questions about the time taken to complete the EORTC QLQ-C30 and QLQ-STO22; the need for help in completing the questionnaires and querying whether any of the questionnaire items were confusing; difficult to answer or upsetting.

OTHER OUTCOMES:
compliance | at the same timepoints when the QoL questionnaires are completed
  Proportion of completed versus expected QoL questionnaires
correlation between QLQ-C30 and STO22 scores | before and after treatment
  correlations between the different established scales of the QLQ-C30 and the hypothesized STO22 scales will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Blazeby, MB, CHB, FRCS, BSc, MD, Study Chair — University Hospitals Bristol and Weston NHS Foundation Trust; Thierry Conroy, MD, Study Chair — Centre Alexis Vautrin
Locations (7):
- Centre Alexis Vautrin, Vandœuvre-lès-Nancy, France
- Germany (2):
  - Universitaetsklinikum Charite, Berlin
  - University of Marburg, Marburg
- Hospital De Navarra, Pamplona, Spain
- Sahlgrenska University Hospital, Gothenburg (Goteborg), Sweden
- United Kingdom (2):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Royal Infirmary, Glasgow, Scotland

REFERENCES:
- [Result] Onate-Ocana LF, Alcantara-Pilar A, Vilar-Compte D, Garcia-Hubard G, Rojas-Castillo E, Alvarado-Aguilar S, Carrillo JF, Blazeby JM, Aiello-Crocifoglio V. Validation of the Mexican Spanish version of the EORTC C30 and STO22 questionnaires for the evaluation of health-related quality of life in patients with gastric cancer. Ann Surg Oncol. 2009 Jan;16(1):88-95. doi: 10.1245/s10434-008-0175-9. Epub 2008 Nov 1. PMID 18979141
- [Result] Sadighi S, Montazeri A, Sedighi Z, Mohagheghi MA, Froutan H. Quality of life in patients with gastric cancer: translation and psychometric evaluation of the Iranian version of EORTC QLQ-STO22. BMC Cancer. 2009 Aug 28;9:305. doi: 10.1186/1471-2407-9-305. PMID 19715606